CLINICAL TRIAL: NCT05152121
Title: The Effect of Fat - Protein Counting on Glycemic Variability in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Additional Insulin for High Fat/Protein in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yasemin Atik Altinok, Dietician PhD, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-12.1/44
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes; Adolescent
Keywords: type 1 diabetes; dietary fat; high energy density meal; glycemic variability
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Qa-SNARE Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- carb counting (Other): Patients using insulin infusion pumps will be placed CGMS for 2 days before starting the study to check whether they are within the target blood glucose levels and normoglycemia will be provided. The content of the first day of the study; The test meal, which is 80 g carbohydrate (29.3%), 70.2 g fat (57.9%), 34.7 g protein (12.7%), will be consumed in the evening meal and normal bolus insulin will be given according to carbohydrate counting. On the second day of the study, instead of the normal bolus for the test meal, the additional insulin for fat-protein by dual wave bolus that.The data obtained will be analyzed by evaluating the CGMS data of all patients by a pediatric endocrinologist experienced in diabetes, CGMS and insulin infusion pump therapy.
  Interventions: Other: Carb and fat counting

INTERVENTIONS:
Other: Carb and fat counting — In the 7 days leading up to the study, participants were contacted to review blood glucose levels with CGMS, food and activity diary. basal rates and insulin carbohydrate ratio and sensitivity factor were changed according to the CGMS values and normoglycemia was achieved.In the study day same meals were served which included high fat, high energy density test meal containing 80 gram carbohydrate (34%), 70 gram fat (66%) and 35 g protein (14%).The participants had to have no glucose fluctuations 2 hours before study entry based on CGMS, no correction boluses for at least 4 hours before the test meal consumption and fasting glycemia in the range of 70-180 mg/dL on both study days.The participants received the test meal calculating insulin dose by CC on the first study day and calculating insulin dose by and fat/protein counting in the second study day. The test meal consumption was completed in 20 minutes under supervision by a caregiver and a dietician of the research team

SUMMARY:
Aim: Dietary carbohydrate is the predominant macronutrient affecting postprandial blood glucose excursions, dietary fat and protein can also significantly impact the postprandial glycemic profile. The aim of this study is to compare the impact of additional dose of extended insulin bolus; using Pankowsko algorithm (PA) to usual standard carbohydrate counting (CC) on postprandial glucose excursions for high fat /high energy density mixed meal for 12 hours.

Methods: In this single-center, non-blinded, randomized, crossover study a high fat, high energy density test meal containing 80 gram carbohydrate (34%), 70 gram fat (66%) and 35 g protein (14%) was given using standard carbohydrate counting (CC) on the first test day and PA was used for the second test day for the same meal. Two methods were compared on postprandial early (0-120 min), late (120-720 min) and total (0-720 min) glucose response in 20 patients with type 1 diabetes mellitus (T1DM), aged 9-18 years on continuous subcutan insulin infusion (CSII) therapy using continuous glucose monitoring system (CGMS).

DETAILED DESCRIPTION:
Children and adolescents with T1DM between the ages of 9-18 and undergoing insulin infusion pump therapy followed in Ege University Pediatric Endocrinology Department will be randomly selected regardless of metabolic control. The selection of the cases will be made from the beginning of the study as the first 30 patients who meet the research participation criteria and agree to participate in the study. Before the research starts, the cases will be told about the application of CGMS, their responsibilities in the research, and an appointment will be given for the insertion of CGMS and this procedure will be applied to all participants. On the day of the appointment, the participant will be put on CGMS, and as long as CGMS is attached, they will be asked to measure capillary blood glucose in their diaries and record them. The subjects will be checked whether they are within the target blood glucose values for 2 days before consuming the test meal and normoglycemia will be provided. On the first day of the study, a test meal with 80 g carbohydrate (29.3%), 70.2 g fat (57.9%), 34.7 g protein (12.7%), will be consumed in the evening meal and carbohydrate counting-normal bolus insulin will be given by administration. On the second day of the study, the additional insulin for fat and protein will be given as a dual wave bolus instead of the normal bolus for the test meal. Then, CGMS will be extracted from the cases, transferred to the computer, and analysis will be made by the researcher, taking into account the capillary blood glucose measurements in the diary.

ELIGIBILITY:
Inclusion Criteria:

1. Children-adolescents with Type 1 DM between the ages of 9-18 and undergoing insulin infusion pump therapy followed by Ege University Faculty of Medicine, Department of Pediatric Endocrine.
2. Those with a body mass index between -2- + 2 SD

Exclusion Criteria:

1. Cases that do not accept to fill in the 'Informed Consent Form'
2. Cases with diseases accompanying T1DM (autoimmune diseases such as celiac, cystic fibrosis, etc.)
3. Body mass index <-2 SD and> +2 SD

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
AUC | AUC was evaluated the day where only carbs were counted and the day were fat and proteins were counted
  The primary outcomes were glucose area under the curve (AUC) and % of time spent in normoglycemia according to CC; PA and modified PA algorithms.

SECONDARY OUTCOMES:
hypoglycemia epizode | Hypoglycemia was evaluated the day where only carbs were counted and the day were fat and proteins were counted
  The secondary outcomes were the number of hypoglycemic events over the study period based on capillary blood glucose measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Darcan, MD Prof, Study Chair — Ege University; Yasemin Atik Altınok, pHD, Principal Investigator — Ege University Fac Of Medicine Department of Pediatrics; Hafize Cetin Işıklar, Nurse, Principal Investigator — Ege University Fac Of Medicine Department of Pediatrics; Gunay Demir, MSci Nurse, Principal Investigator — Ege University Fac Of Medicine Department of Pediatrics; Samim Ozen, MD,PhD, Principal Investigator — Ege University Fac Of Medicine Department of Pediatrics
Locations (1):
- Ege University Faculty of Medicine Department of Pediatrics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Gingras V, Bonato L, Messier V, Roy-Fleming A, Smaoui MR, Ladouceur M, Rabasa-Lhoret R. Impact of macronutrient content of meals on postprandial glucose control in the context of closed-loop insulin delivery: A randomized cross-over study. Diabetes Obes Metab. 2018 Nov;20(11):2695-2699. doi: 10.1111/dom.13445. Epub 2018 Jul 18. PMID 29931719
- [Background] American Diabetes Association. 5. Facilitating Behavior Change and Well-being to Improve Health Outcomes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S53-S72. doi: 10.2337/dc21-S005. PMID 33298416
- [Background] Smart CE, Annan F, Higgins LA, Jelleryd E, Lopez M, Acerini CL. ISPAD Clinical Practice Consensus Guidelines 2018: Nutritional management in children and adolescents with diabetes. Pediatr Diabetes. 2018 Oct;19 Suppl 27:136-154. doi: 10.1111/pedi.12738. No abstract available. PMID 30062718
- [Background] Pankowska E, Szypowska A, Lipka M, Szpotanska M, Blazik M, Groele L. Application of novel dual wave meal bolus and its impact on glycated hemoglobin A1c level in children with type 1 diabetes. Pediatr Diabetes. 2009 Aug;10(5):298-303. doi: 10.1111/j.1399-5448.2008.00471.x. Epub 2008 Oct 20. PMID 19175902
- [Background] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583
- [Background] Bell KJ, Smart CE, Steil GM, Brand-Miller JC, King B, Wolpert HA. Impact of fat, protein, and glycemic index on postprandial glucose control in type 1 diabetes: implications for intensive diabetes management in the continuous glucose monitoring era. Diabetes Care. 2015 Jun;38(6):1008-15. doi: 10.2337/dc15-0100. PMID 25998293
- [Result] Jones SM, Quarry JL, Caldwell-McMillan M, Mauger DT, Gabbay RA. Optimal insulin pump dosing and postprandial glycemia following a pizza meal using the continuous glucose monitoring system. Diabetes Technol Ther. 2005 Apr;7(2):233-40. doi: 10.1089/dia.2005.7.233. PMID 15857224
- [Result] Wolever TM, Mullan YM. Sugars and fat have different effects on postprandial glucose responses in normal and type 1 diabetic subjects. Nutr Metab Cardiovasc Dis. 2011 Sep;21(9):719-25. doi: 10.1016/j.numecd.2010.12.005. Epub 2011 Feb 16. PMID 21330118
- [Result] Pankowska E, Blazik M, Groele L. Does the fat-protein meal increase postprandial glucose level in type 1 diabetes patients on insulin pump: the conclusion of a randomized study. Diabetes Technol Ther. 2012 Jan;14(1):16-22. doi: 10.1089/dia.2011.0083. Epub 2011 Oct 20. PMID 22013887
- [Result] Smart CE, Evans M, O'Connell SM, McElduff P, Lopez PE, Jones TW, Davis EA, King BR. Both dietary protein and fat increase postprandial glucose excursions in children with type 1 diabetes, and the effect is additive. Diabetes Care. 2013 Dec;36(12):3897-902. doi: 10.2337/dc13-1195. Epub 2013 Oct 29. PMID 24170749
- [Result] Wolpert HA, Atakov-Castillo A, Smith SA, Steil GM. Dietary fat acutely increases glucose concentrations and insulin requirements in patients with type 1 diabetes: implications for carbohydrate-based bolus dose calculation and intensive diabetes management. Diabetes Care. 2013 Apr;36(4):810-6. doi: 10.2337/dc12-0092. Epub 2012 Nov 27. PMID 23193216
- [Result] Paterson MA, Smart CEM, Lopez PE, Howley P, McElduff P, Attia J, Morbey C, King BR. Increasing the protein quantity in a meal results in dose-dependent effects on postprandial glucose levels in individuals with Type 1 diabetes mellitus. Diabet Med. 2017 Jun;34(6):851-854. doi: 10.1111/dme.13347. Epub 2017 Mar 19. PMID 28257160
- [Result] van der Hoogt M, van Dyk JC, Dolman RC, Pieters M. Protein and fat meal content increase insulin requirement in children with type 1 diabetes - Role of duration of diabetes. J Clin Transl Endocrinol. 2017 Oct 10;10:15-21. doi: 10.1016/j.jcte.2017.10.002. eCollection 2017 Dec. PMID 29204367
- [Result] Neu A, Behret F, Braun R, Herrlich S, Liebrich F, Loesch-Binder M, Schneider A, Schweizer R. Higher glucose concentrations following protein- and fat-rich meals - the Tuebingen Grill Study: a pilot study in adolescents with type 1 diabetes. Pediatr Diabetes. 2015 Dec;16(8):587-91. doi: 10.1111/pedi.12224. Epub 2014 Oct 20. PMID 25330823
- [Result] Paterson MA, Smart CE, Lopez PE, McElduff P, Attia J, Morbey C, King BR. Influence of dietary protein on postprandial blood glucose levels in individuals with Type 1 diabetes mellitus using intensive insulin therapy. Diabet Med. 2016 May;33(5):592-8. doi: 10.1111/dme.13011. Epub 2015 Dec 6. PMID 26499756
- [Result] Evans M, Smart CEM, Paramalingam N, Smith GJ, Jones TW, King BR, Davis EA. Dietary protein affects both the dose and pattern of insulin delivery required to achieve postprandial euglycaemia in Type 1 diabetes: a randomized trial. Diabet Med. 2019 Apr;36(4):499-504. doi: 10.1111/dme.13875. Epub 2019 Feb 20. PMID 30537305
- [Result] Lopez PE, Evans M, King BR, Jones TW, Bell K, McElduff P, Davis EA, Smart CE. A randomized comparison of three prandial insulin dosing algorithms for children and adolescents with Type 1 diabetes. Diabet Med. 2018 Oct;35(10):1440-1447. doi: 10.1111/dme.13703. Epub 2018 Jun 19. PMID 29873107
- [Result] Kordonouri O, Hartmann R, Remus K, Blasig S, Sadeghian E, Danne T. Benefit of supplementary fat plus protein counting as compared with conventional carbohydrate counting for insulin bolus calculation in children with pump therapy. Pediatr Diabetes. 2012 Nov;13(7):540-4. doi: 10.1111/j.1399-5448.2012.00880.x. Epub 2012 Jul 6. PMID 22765260